CLINICAL TRIAL: NCT02600533
Title: Increasing Minority Group Participation in Clinical Trials a Randomized Controlled Study of an Office-based Educational Video
Brief Title: Increasing Minority Participation in Clinical Trials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Meharry-Vanderbilt Alliance (Other)
Responsible Party: Principal Investigator, Consuelo H Wilkins, Executive Director of the Meharry-Vanderbilt Alliance, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14117; P30CA068485 (NIH)
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Clinical Trial
Keywords: minority group recruitment; stages of implementation; clinical trials education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care/control group (No Intervention): First, participants will complete a brief electronic survey measuring their opinions on clinical trials. Next, participants in the standard of care group will be provided standard educational resources (booklet and DVD), with no additional instructions. Participants in this groups will be informed that a team member will call him/her in approximately 1 week to ask him/her the (same) questions about clinical research.
- Video viewing group (Experimental): First, participants will complete a brief electronic survey measuring their opinions on clinical trials. Next, participants in the video viewing group will watch the 10-minute DVD video on tablet devices using headphones in the clinic. Participants in this groups will be informed that a team member will call him/her in approximately 1 week to ask him/her the (same) questions about clinical research.
  Interventions: Procedure: Video viewing group

INTERVENTIONS:
Procedure: Video viewing group — First, participants will complete a brief electronic survey measuring their opinions on clinical trials. Next, participants in the video viewing group will watch the 10-minute DVD video on tablet devices using headphones in the clinic. Participants in this groups will be informed that a team member will call him/her in approximately 1 week to ask him/her the (same) questions about clinical research.
  Other Names: video group
  Arms: Video viewing group

SUMMARY:
This study will measure the effects of an office-based, clinical trial education video on clinical trial knowledge and enrollment in clinical trials, in a clinical sample with no previous history of clinical trial participation. This study will also determine the feasibility of implementing an office-based video educational program.

DETAILED DESCRIPTION:
Clinical trials are essential to scientific discovery and are critical to translating research in to practice. Despite their significance, clinical trial participation rates remain low, especially among underrepresented minority groups. Several barriers exist to minority group participation in clinical trial, one of which lack of awareness about clinical trials. Video educational programs show promise as an effective strategy to increase knowledge and clinical trial participation. The specific aims are as follows:

1. Measure the effects of an office-based, clinical trial education video on clinical trial knowledge and enrollment in clinical trials, in a clinical sample with no previous history of clinical trial participation.
2. Determine the feasibility of implementing an office-based video educational program.

ELIGIBILITY:
Inclusion Criteria:

Participants will be patients of Vanderbilt-Ingram Cancer Center (VICC) with a diagnosis of cancer Participants will have no previous history of clinical trial research participation

Exclusion Criteria:

* Previous history of clinical trial research participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
study feasibility | 12 months
  The stages of implementation completion (SIC) measure will be used as an internal tool utilized by the study team to track time to achievement of key implementation milestones. An 8-stage implementation plan to measure feasibility of the office-based educational program will be executed across 3 phases. Three scores will be derived from the SIC measure. The first score is the number of stages completed. The second score is the time spent at each stage. The third score is the proportion of activities completed at each stage. Implementation of the SIC model poses no additional burden on study participants.

SECONDARY OUTCOMES:
Clinical trial participation | 12 months
  Information on clinical trial participation will be collected by a team member by reviewing the participants' health record and by contacting the VICC clinical trial team.
Clinical trial knowledge survey | 7-10 days
  This survey consist of 22-items assessing a participants views on clinical trials on 5 domains (positive beliefs, safety, information needs, negative expectations, and patient involvement).
Likelihood to participate survey | 7-10 days
  This survey consist of 5-items assessing reasons for not participating in research, views about sources of research, views about sharing of research data, trust, and willingness to advise research teams.

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo H. Wilkins, MD, Principal Investigator — Meharry-Vanderbilt Alliance, Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Ingram Cancer Center, Vanderbilt University Medical Center, Nashville, Tennessee, United States